CLINICAL TRIAL: NCT06914115
Title: Effect of Transcutaneous Auricular Nerve Stimulation vs Body Rocking Exercises on Spasticity of Upper Limb in Young Stroke Patients
Brief Title: Effect of Transcutaneous Auricular Nerve Stimulation vs Body Rocking Exercises on Spasticity of Upper Limb
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/816
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Spasticity, Muscle
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TANS Group (Experimental)
  Interventions: Combination Product: TANS Group
- Body Rocking Exercise (Experimental)
  Interventions: Combination Product: Body Rocking Exercise

INTERVENTIONS:
Combination Product: TANS Group — The TANS Group will receive low-frequency electrical stimulation (20-30 Hz) via a TENS device on the auricular vagus nerve for 30 minutes, 3-4 times per week for 8 weeks. This non-invasive therapy aims to reduce spasticity, enhance neuroplasticity, and improve motor function and independence, assessed through standardized scales.
  Arms: TANS Group
Combination Product: Body Rocking Exercise — Group 2: Body Rocking Exercise Group Participants will perform rhythmic body rocking exercises for 20-30 minutes, 3-4 times per week for 8 weeks to reduce spasticity and improve motor coordination. Group 3: Control Group (Usual Rehabilitation) Participants will receive standard stroke rehabilitation (therapy, stretching, functional training) for 20-30 minutes, 3-4 times per week for 8 weeks as a baseline comparison.
  Arms: Body Rocking Exercise

SUMMARY:
The primary aim of this study is to compare the effect of TANS and body rocking exercises on reducing upper limb spasticity in young stroke patients( under 50). Specific objectives include evaluating changes in muscle tone, motor function, pain reduction, and functional independence following each intervention.

DETAILED DESCRIPTION:
This randomized controlled trial, RCT, will involve 42 young stroke patients with upper limb spasticity randomly assigned to three groups, transcutaneous auricular nerve stimulation, body rocking exercise, or control group, usually rehabilitation. Participants will receive 30-minute transcutaneous nerve stimulation session or 20 to 30-minute body rocking exercise in session 3 to 4 times a week over an 8-week period. Key outcome measures include the Modified Ashworth Scale for Spasticity, the Fusel-Meyer Assessment for Motor Function, the Numeric Rating Scale for Pain, and Stroke Impact Scale for Functional Independence.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-50 years
* Diagnosed with stroke (ischemic or hemorrhagic)
* Upper limb spasticity (Modified Ashworth Scale score ≥1)
* Post-stroke duration of ≥3 months
* Able to follow verbal and physical instructions
* No contraindications to electrical stimulation or exercise therapy

Exclusion Criteria:

* Severe cognitive impairment or communication disorders
* History of epilepsy or uncontrolled seizures
* Pacemaker or implanted medical devices
* Severe cardiac, orthopedic, or neurological conditions
* Uncontrolled hypertension or diabetes
* Participation in another spasticity-related trial

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | 12 Months
  Assesses spasticity (0 = no increase, 4 = rigid limb).
Fugl-Meyer Assessment (FMA) | 12 Months
  Evaluates motor function (0-66, higher = better function).
Numeric Rating Scale (NRS) | 12 Months
  Measures pain (0 = no pain, 10 = severe pain).

CONTACTS AND LOCATIONS:
Locations (1):
- City Rehabilitation Center, Okāra, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No